CLINICAL TRIAL: NCT06487910
Title: Pilot Study on the Design of a 3D-printed Differential Pressure Distribution Orthosis for the Treatment of Post-burn Hypertrophic Scarring
Brief Title: Differential Pressure Distribution Orthosis by 3D Printing Process in the Treatment of Post-burn Hypertrophic Scarring
Acronym: EPIDERM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-01-CHRMT
Record Dates: First submitted 2024-06-19; First posted 2024-07-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Burns; Hypertrophic Scar
MeSH Terms: conditions — Burns; Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D scan measurment (Experimental): patients included in the study will undergo a 3D scan measurement of on or more burn scars. This measurement will then be digitally modified in preparation for the manufacture of the "differential pressure distribution orthosis". The orthosis will then be manufactured using a 3D printing process.
  Interventions: Device: 3D scan measurment

INTERVENTIONS:
Device: 3D scan measurment — patients included in the study will undergo a 3D scan measurement of on or more burn scars. This measurement will then be digitally modified in preparation for the manufacture of the "differential pressure distribution orthosis". The orthosis will then be manufactured using a 3D printing process.

SUMMARY:
This is a pilot, single-center, feasibility study to evaluate a new 3D printing method for ORDP design.

To our knowledge, there is no technical or clinical evaluation of ORDPs, particularly in the treatment of hypertrophic scars. The aim of our study is therefore to assess the feasibility of an innovative method of designing ORDPs for the curative treatment of post-burn hypertrophic scars, using a 3D printing process, and to describe the procedures (production time and cost).

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients aged > 18 years old
* Patient with at least one hypertrophic burn scar in the process of healing localized on a skin area that can benefit from a compression garment and requiring the use of an ORDP
* Patient able to give informed consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patients under guardianship, curatorship or safeguard of justice
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Sucess of the manufacture process of the orthosis | 2 to 3 hours after inclusion
  Defined as the compliance with all three of the following specifications: 1) oval shapes are approximately 2 mm thick, 2) absence of wounding areas (prickly or sharp), 3) a satisfactory morphological match with the area to be treated.

SECONDARY OUTCOMES:
Time of conception | 2 to 3 hours after inclusion
  Total time to make the orthosis (minutes)
Total time to design the orthosis | 2 to 3 hours after inclusion
  Total time to design the orthosis (minutes)
Total cost of the orthosis fabrication | 2 to 3 hours after inclusion
  Total cost of the orthosis fabrication (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Loic BANASZAK, Principal Investigator — CHR Metz Thionville Hopital Félix Maréchal
Locations (1):
- CHR Metz-Thionville/Hopital Félix Maréchal, Metz, France

IPD SHARING:
Plan to Share IPD: No